CLINICAL TRIAL: NCT02666157
Title: Comparison of Efficacy and Safety Among DAbigatran, RIvaroxaban, and ApixabaN in Patients HavinG Non-Valvular Atrial Fibrillation in Taiwan (DARING-AF Study)
Brief Title: Comparison of Efficacy and Safety Among Dabigatran, Rivaroxaban, and Apixaban in Non-Valvular Atrial Fibrillation
Acronym: DARING-AF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cheng-Kung University Hospital (Other)
Collaborators: Tainan Municipal Hospital (Other); E-DA Hospital (Other); National Cheng-Kung University Hospital Dou-Liou Branch (Unknown); Ministry of Health and Welfare, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A-BR-104-049
Record Dates: First submitted 2016-01-24; First posted 2016-01-28 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; stroke; systemic embolism; bleeding; oral anticoagulant
MeSH Terms: conditions — Atrial Fibrillation; Stroke; Hemorrhage | interventions — Dabigatran; Rivaroxaban; apixaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dabigatran (Active Comparator): oral dabigatran etexilate capsule 110 or 150 mg (110 mg in specific population) bid for entire study period
  Interventions: Drug: Dabigatran etexilate
- Rivaroxaban (Active Comparator): oral rivaroxaban film-coated tablet 15 or 20 mg (10 or 15 mg in specific population) qd for entire study period
  Interventions: Drug: Rivaroxaban
- Apixaban (Active Comparator): oral apixaban 5 mg (2.5 mg in specific population) bid for entire study period
  Interventions: Drug: Apixaban

INTERVENTIONS:
Drug: Dabigatran etexilate — this drug is administered twice per day for the entire study period
  Other Names: Pradaxa
  Arms: Dabigatran
Drug: Rivaroxaban — this drug is administered once per day for the entire study period
  Other Names: Xarelto
  Arms: Rivaroxaban
Drug: Apixaban — this drug is administered twice per day for the entire study period
  Other Names: Eliquis
  Arms: Apixaban

SUMMARY:
1. The recent development of novel oral anticoagulants (NOACs), including direct thrombin inhibitor (dabigatran) and factor Xa inhibitors (rivaroxaban, apixaban, and edoxaban), could potentially overcome many drawbacks of warfarin, and might provide a safer, and even more effective and convenient alternative approach to warfarin in non-valvular atrial fibrillation (NVAF), especially in Asians.
2. According to the results of a meta-analysis comparing Asians and non-Asians, NOACs are preferentially indicated in Asians in terms of both efficacy and safety.
3. There is no randomized controlled trial with sufficient power to directly compare the efficacy and safety among NOACs in NVAF, not to speak of Asians and Chinese.
4. Indirect comparisons are only based on observation with a lot of limitations such as heterogeneous background characteristics, difference in study design, and diversity in time within therapeutic range in control group. The findings from indirect comparisons are not conclusive but only hypothesis-generating.
5. This investigator-initiated prospective randomized open blinded end-point clinical trial will directly compare the efficacy and safety among 3 NOACs in patients with NVAF in Taiwan. We hypothesize that rivaroxaban or apixaban is non-inferior to dabigatran in terms of the efficacy.

DETAILED DESCRIPTION:
1. participants

   a. eligible participants are randomly assigned to dabigatran, rivaroxaban, or apixaban with allocation ratio of 1:1:1
   * Patients are randomly assigned to receive dabigatran (110 or 150 mg twice daily), rivaroxaban (15 or 20 mg daily), or apixaban (5 mg twice daily) with dosage and frequency approved by the Ministry of Health and Welfare, Taiwan. Reduced doses (dabigatran 110 mg twice daily, rivaroxaban 10 or 15 mg daily, or apixaban 2.5 mg twice daily) are allowed in a subset of patients with one or more of the following criteria: an age of at least 80 years, a body weight of no more than 60 kg, a serum creatinine level ≥1.5 mg per deciliter (133 μmol per liter) or creatinine clearance around 30 to 49 ml per minute)
2. blood sampling, genotyping, and measurement of biomarkers

   a. bood samples (13 mL) from peripheral veins in all study subjects at baseline and 10 mL 3 months later, and stored for enzyme-linked immunosorbent assay as well as genotyping
3. outcome follow-up a. clinical follow-up is performed and clinical outcomes are obtained by clinic visit, telephone call or direct contact with participants or subjects' family quarterly after treatment for 2 times, then every 6 months

ELIGIBILITY:
Inclusion Criteria: Known AF (paroxysmal or persistent/ permanent) who are suitable and ready for NOAC treatment plus at least one of the following criteria

* Prior ischemic stroke, transient ischemic accident or systemic embolism
* Left ventricular ejection fraction ≤40% (documented by echocardiography or contrast ventriculography)
* Symptomatic congestive heart failure (≥ New York Heart Association Functional Class 2) within 6 months before screening
* Age ≥75 years
* Age ≥65 but <75 years with diabetes mellitus, hypertension or coronary artery disease

Exclusion Criteria: Subjects are excluded if they have at least one of the following situations before screening:

* Known severe (i.e. hemodynamically significant) mitral stenosis regardless of having received operation
* Time elapsed from the onset of stroke ≤7 days
* Bleeding tendency
* Creatinine clearance rate ≤30 mL/min
* Known active liver disease (persistent elevation of alanine aminotransferase, aspartate transaminase or alkaline phosphatase ≥3 × upper normal limit; or advanced liver cirrhosis ≥Pugh B)
* Pregnancy
* Recent documented active malignancy or radiation therapy (≤6 months) and not expected to survive 3 years
* Unwilling to give informed consent
* Conditions other than AF that required anticoagulation
* Anemia (hemoglobin level <90 g/L) or thrombocytopenia (platelet count <100 × 109/L)
* Persistent uncontrolled hypertension (systolic blood pressure >180 mmHg or diastolic blood pressure >100 mmHg)
* Active infective endocarditis
* Patients considered unreliable by the investigator or have a life expectancy less than the expected duration of the trial because of concomitant disease, or has any condition which in the opinion of the investigator, would not allow safe participation in the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3672 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Time to the occurrence of the major embolic events | up to 36 months
  a composite of stroke (ischemic or hemorrhagic), transient ischemic attack or systemic embolism

SECONDARY OUTCOMES:
Time to the occurrence of the major embolic events and death | up to 36 months
  a composite of all stroke (including hemorrhagic), systemic embolism, and death
Time to the occurrence of the major embolic and vascular events | up to 36 months
  a composite of all stroke, systemic embolism, pulmonary embolism, acute myocardial infarction, and vascular death
Time to the occurrence of all clinically relevant bleeding events | up to 36 months
  a composite of major bleeding or clinically relevant non-major bleeding events

OTHER OUTCOMES:
Time to the occurrence of all stroke | up to 36 months
  stroke is defined as a focal loss of neurological function caused by an ischemic or hemorrhagic event with residual symptoms at least 24 hours after onset or leading to death
Time to the occurrence of systemic embolism | up to 36 months
  embolic events excluding stroke, pulmonary embolism or venous thromboembolism
Time to the occurrence of transient ischemic attack | up to 36 months
  a transient focal loss of neurological function caused by an ischemic event with complete recovery within 24 hours after onset
Time to the occurrence of death | up to 36 months
  all-cause death includes vascular and non-vascular causes
Time to the occurrence of pulmonary embolism | up to 36 months
  clinical diagnosis of pulmonary embolism should be confirmed by an image study
Time to the occurrence of acute myocardial infarction | up to 36 months
  acute myocardial infarction is defined in accordance with the universal definition proposed in 2012
Time to the occurrence of vascular death | up to 36 months
  sudden cardiac death, fatal stroke, fatal myocardial infarction, any other death for which there is no clearly documented non-vascular cause, and death from bleeding
Time to the occurrence of hospitalization for congestive heart failure | up to 36 months
  decompensated congestive heart failure requiring hospitalization for stabilization
Time to the occurrence of advanced chronic kidney disease | up to 36 months
  defined as estimated glomerular filtration rate <30 mL/min/1.73m2 confirmed by 2 separate laboratory tests within 3 months
Time to the occurrence of cardiogenic shock | up to 36 months
  symptoms and signs of organ hypoperfusion (e.g. cool peripheries, oliguria) plus one of the following parameters: systolic blood pressure 90 mmHg or less, hypotension requiring inotropic/vasopressor therapy remaining after fluid challenge, heart rate of at least 60 bpm, or a cardiac index of 2.2 L/min/m2 or less
Time to the occurrence of any revascularization for peripheral artery disease | up to 36 months
  percutaneous transluminal angioplasty or bypass surgery for low extremity artery disease
Time to the occurrence of any revascularization for coronary artery disease | up to 36 months
  percutaneous coronary intervention or coronary artery bypass grafting for obstructive coronary artery disease
Time to occurrence of any revascularization for carotid or vertebral artery stenosis | up to 36 months
  endovascular therapy, endarterectomy or bypass surgery for carotid or vertebral artery stenosis
Time to the occurrence of major bleeding events | up to 36 months
  defined as bleeding to cause a drop in hemoglobin level >= 2g/dL, fatal bleeding, life-threatening bleeding, or symptomatic bleeding at critical sites (including intracranial, retroperitoneal, intraocular, or intrapericardial)
Time to the occurrence of life-threatening bleeding events | up to 36 months
  defined as fatal bleeding, symptomatic intracranial hemorrhage, bleeding to cause a drop in hemoglobin level >=5g/dL, bleeding requiring transfusion with >=4u blood component, bleeding requiring vasopressor administration, or bleeding needing surgery for hemostasis
Time to the occurrence of minor bleeding events | up to 36 months
  non-major or non-life-threatening bleeding events
Time to the occurrence of clinically relevant non-major bleeding events | up to 36 months
  clinically overt bleeding that does not satisfy the criteria for major bleeding and that leads to hospital admission, physician-guided medical or surgical treatment, or a change in antithrombotic therapy
Time to the occurrence of major or minor bleeding events | up to 36 months
  major or minor bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Ting-Hsing Chao, MD, Study Chair — National Cheng-Kung University Hospital
Locations (5):
- Taiwan (5):
  - National Cheng Kung University Hospital, Tainan, Tainan City
  - Tainan Hospital Ministry of Health and Welfare, Tainan, Tainan City
  - National Cheng Kung University Hospital Dou-Liou Branch, Dou-Liou City
  - E-DA Hospital, Kaohsiung City
  - Tainan Municipal Hospital, Tainan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chiang CE, Zhang S, Tse HF, Teo WS, Omar R, Sriratanasathavorn C. Atrial fibrillation management in Asia: from the Asian expert forum on atrial fibrillation. Int J Cardiol. 2013 Mar 20;164(1):21-32. doi: 10.1016/j.ijcard.2011.12.033. Epub 2012 Jan 10. PMID 22240753
- [Background] Chiang CE, Wang KL, Lip GY. Stroke prevention in atrial fibrillation: an Asian perspective. Thromb Haemost. 2014 May 5;111(5):789-97. doi: 10.1160/TH13-11-0948. Epub 2014 Feb 6. PMID 24500243
- [Background] Lin LJ, Cheng MH, Lee CH, Wung DC, Cheng CL, Kao Yang YH. Compliance with antithrombotic prescribing guidelines for patients with atrial fibrillation--a nationwide descriptive study in Taiwan. Clin Ther. 2008 Sep;30(9):1726-36. doi: 10.1016/j.clinthera.2008.09.010. PMID 18840379
- [Background] Chang CH, Yang YH, Chen JH, Lin LJ. Cost-effectiveness of dabigatran etexilate for the prevention of stroke and systemic embolism in atrial fibrillation in Taiwan. Thromb Res. 2014 May;133(5):782-9. doi: 10.1016/j.thromres.2014.02.024. Epub 2014 Mar 3. PMID 24642004
- [Background] Lip GY, Wang KL, Chiang CE. Non-vitamin K antagonist oral anticoagulants (NOACs) for stroke prevention in Asian patients with atrial fibrillation: time for a reappraisal. Int J Cardiol. 2015 Feb 1;180:246-54. doi: 10.1016/j.ijcard.2014.11.182. Epub 2014 Nov 26. PMID 25463377
- [Background] Connolly SJ, Ezekowitz MD, Yusuf S, Eikelboom J, Oldgren J, Parekh A, Pogue J, Reilly PA, Themeles E, Varrone J, Wang S, Alings M, Xavier D, Zhu J, Diaz R, Lewis BS, Darius H, Diener HC, Joyner CD, Wallentin L; RE-LY Steering Committee and Investigators. Dabigatran versus warfarin in patients with atrial fibrillation. N Engl J Med. 2009 Sep 17;361(12):1139-51. doi: 10.1056/NEJMoa0905561. Epub 2009 Aug 30. PMID 19717844
- [Background] Patel MR, Mahaffey KW, Garg J, Pan G, Singer DE, Hacke W, Breithardt G, Halperin JL, Hankey GJ, Piccini JP, Becker RC, Nessel CC, Paolini JF, Berkowitz SD, Fox KA, Califf RM; ROCKET AF Investigators. Rivaroxaban versus warfarin in nonvalvular atrial fibrillation. N Engl J Med. 2011 Sep 8;365(10):883-91. doi: 10.1056/NEJMoa1009638. Epub 2011 Aug 10. PMID 21830957
- [Background] Granger CB, Alexander JH, McMurray JJ, Lopes RD, Hylek EM, Hanna M, Al-Khalidi HR, Ansell J, Atar D, Avezum A, Bahit MC, Diaz R, Easton JD, Ezekowitz JA, Flaker G, Garcia D, Geraldes M, Gersh BJ, Golitsyn S, Goto S, Hermosillo AG, Hohnloser SH, Horowitz J, Mohan P, Jansky P, Lewis BS, Lopez-Sendon JL, Pais P, Parkhomenko A, Verheugt FW, Zhu J, Wallentin L; ARISTOTLE Committees and Investigators. Apixaban versus warfarin in patients with atrial fibrillation. N Engl J Med. 2011 Sep 15;365(11):981-92. doi: 10.1056/NEJMoa1107039. Epub 2011 Aug 27. PMID 21870978
- [Background] Giugliano RP, Ruff CT, Braunwald E, Murphy SA, Wiviott SD, Halperin JL, Waldo AL, Ezekowitz MD, Weitz JI, Spinar J, Ruzyllo W, Ruda M, Koretsune Y, Betcher J, Shi M, Grip LT, Patel SP, Patel I, Hanyok JJ, Mercuri M, Antman EM; ENGAGE AF-TIMI 48 Investigators. Edoxaban versus warfarin in patients with atrial fibrillation. N Engl J Med. 2013 Nov 28;369(22):2093-104. doi: 10.1056/NEJMoa1310907. Epub 2013 Nov 19. PMID 24251359
- [Background] Hori M, Connolly SJ, Zhu J, Liu LS, Lau CP, Pais P, Xavier D, Kim SS, Omar R, Dans AL, Tan RS, Chen JH, Tanomsup S, Watanabe M, Koyanagi M, Ezekowitz MD, Reilly PA, Wallentin L, Yusuf S; RE-LY Investigators. Dabigatran versus warfarin: effects on ischemic and hemorrhagic strokes and bleeding in Asians and non-Asians with atrial fibrillation. Stroke. 2013 Jul;44(7):1891-6. doi: 10.1161/STROKEAHA.113.000990. Epub 2013 Jun 6. PMID 23743976
- [Background] Ruff CT, Giugliano RP, Braunwald E, Hoffman EB, Deenadayalu N, Ezekowitz MD, Camm AJ, Weitz JI, Lewis BS, Parkhomenko A, Yamashita T, Antman EM. Comparison of the efficacy and safety of new oral anticoagulants with warfarin in patients with atrial fibrillation: a meta-analysis of randomised trials. Lancet. 2014 Mar 15;383(9921):955-62. doi: 10.1016/S0140-6736(13)62343-0. Epub 2013 Dec 4. PMID 24315724
- [Background] Lip GY, Larsen TB, Skjoth F, Rasmussen LH. Indirect comparisons of new oral anticoagulant drugs for efficacy and safety when used for stroke prevention in atrial fibrillation. J Am Coll Cardiol. 2012 Aug 21;60(8):738-46. doi: 10.1016/j.jacc.2012.03.019. Epub 2012 May 9. PMID 22575324
- [Background] Ezekowitz MD, Connolly S, Parekh A, Reilly PA, Varrone J, Wang S, Oldgren J, Themeles E, Wallentin L, Yusuf S. Rationale and design of RE-LY: randomized evaluation of long-term anticoagulant therapy, warfarin, compared with dabigatran. Am Heart J. 2009 May;157(5):805-10, 810.e1-2. doi: 10.1016/j.ahj.2009.02.005. PMID 19376304
- [Background] ROCKET AF Study Investigators. Rivaroxaban-once daily, oral, direct factor Xa inhibition compared with vitamin K antagonism for prevention of stroke and Embolism Trial in Atrial Fibrillation: rationale and design of the ROCKET AF study. Am Heart J. 2010 Mar;159(3):340-347.e1. doi: 10.1016/j.ahj.2009.11.025. PMID 20211293
- [Background] Lopes RD, Alexander JH, Al-Khatib SM, Ansell J, Diaz R, Easton JD, Gersh BJ, Granger CB, Hanna M, Horowitz J, Hylek EM, McMurray JJ, Verheugt FW, Wallentin L; ARISTOTLE Investigators. Apixaban for reduction in stroke and other ThromboemboLic events in atrial fibrillation (ARISTOTLE) trial: design and rationale. Am Heart J. 2010 Mar;159(3):331-9. doi: 10.1016/j.ahj.2009.07.035. PMID 20211292
- [Background] Ruff CT, Giugliano RP, Antman EM, Crugnale SE, Bocanegra T, Mercuri M, Hanyok J, Patel I, Shi M, Salazar D, McCabe CH, Braunwald E. Evaluation of the novel factor Xa inhibitor edoxaban compared with warfarin in patients with atrial fibrillation: design and rationale for the Effective aNticoaGulation with factor xA next GEneration in Atrial Fibrillation-Thrombolysis In Myocardial Infarction study 48 (ENGAGE AF-TIMI 48). Am Heart J. 2010 Oct;160(4):635-41. doi: 10.1016/j.ahj.2010.06.042. PMID 20934556
- [Background] Wang KL, Lip GY, Lin SJ, Chiang CE. Non-Vitamin K Antagonist Oral Anticoagulants for Stroke Prevention in Asian Patients With Nonvalvular Atrial Fibrillation: Meta-Analysis. Stroke. 2015 Sep;46(9):2555-61. doi: 10.1161/STROKEAHA.115.009947. Epub 2015 Jul 30. PMID 26304863